CLINICAL TRIAL: NCT01741012
Title: Phase I, Safety and Immunogenicity of Gardasil® in Systemic Lupus Erythematosus.
Brief Title: Study to Determine if Gardasil Vaccine is Safe and Effective in Lupus Patients
Acronym: GARDASIL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Patricia Dhar, Assistant Professor of Medicine, Wayne State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0412GARDASIL
Record Dates: First submitted 2012-11-14; First posted 2012-12-04 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gardasil (Experimental): 0.5 ml single dose Gardasil vaccine given at three separate visits
  Interventions: Drug: Gardasil

INTERVENTIONS:
Drug: Gardasil — 0.5 ml Gardasil vaccine in single dose prefilled syringes at Visit 2, Visit 4 and Visit 6

SUMMARY:
Cervical neoplasia is increased in women with SLE most likely due to cervical infection with human papilloma virus (HPV). 70% of cervical cancer is caused by HPV types 16 and 18. Gardasil vaccine prevents cervical infection with HPV types 16 and 18. Thus lupus patients (who are susceptible to cervical cancer) may benefit from getting Gardasil vaccine which can prevent cervical cancer. Vaccines are generally safe and efficacious in SLE but no studies have been done on the use of this vaccine in SLE. The investigators hypothesize that Gardasil vaccine is safe and effective in SLE. This study will look at vaccine safety in patients with mild to moderate and minimally active or inactive SLE and measure how well they make protective antibodies after receiving the vaccine. In other words this will check how well the vaccine works in SLE.

DETAILED DESCRIPTION:
To gather safety information and adverse events on the use of Gardasil® in mild to moderate and minimally active or inactive SLE.

To gather information on SLE disease activity flares after vaccination with Gardasil®.

To gather information on the immunogenicity or development of protective anti HPV antibodies SLE after vaccination with Gardasil®.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of systemic lupus erythematosis (SLE) by the American College of Rheumatology (ACR) Criteria.

History of a positive antinuclear antibody (ANA) test result at any time in the past.

40 participants with history of mild to moderate SLE disease Minimally active or inactive SLE disease, i.e., (Safety of Estrogens in Lupus Erythematosis National Assessment (SELENA) Systemic Lupus Erythematosus Disease Activity Index (SLEDAI), SELENA-SLEDAI ≤2 at the start of the study.

Age ≥ 18 years and ≤ 50 years. Gender: females Ability to provide informed consent. Maintenance Prednisone dose ≤ 15 mg/day. Plaquenil ≤ 400 mg/day.

Exclusion Criteria:

Hypersensitivity to any vaccine component Active infections including but not limited to human immunodeficiency virus (HIV positive), Hepatitis B or C, tuberculosis.

Positive purified protein derivative (PPD) test results without evidence of prior treatment or administration of bacilli Calmette-Guerin (BCG) vaccine. A positive PPD is defined as ≥ 5 mm induration 24-38 hours after receiving 5TU (TU=tuberculin units) of PPD.

Pregnancy or desire to become pregnant during the study period. Breast feeding. Inability to complete the immunization series. Received any blood product or component in the previous 6 months before enrollment.

Received any inactivated vaccine product within 14 days before enrollment. Received any live vaccine product within 21 days before enrollment.

Fever (temperature > 100°F) at the time of enrollment. Inability to provided informed consent.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia J Dhar, MD, Principal Investigator — Wayne State University
Locations (1):
- DCaTS-Clinical Research Center, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared with any researcher, only aggregated de-identified data

REFERENCES:
- [Derived] Dhar JP, Essenmacher L, Dhar R, Magee A, Ager J, Sokol RJ. The safety and immunogenicity of Quadrivalent HPV (qHPV) vaccine in systemic lupus erythematosus. Vaccine. 2017 May 9;35(20):2642-2646. doi: 10.1016/j.vaccine.2017.04.001. Epub 2017 Apr 9. PMID 28404357
- See also: Clinical Research Services Center, Wayne State University School of Medicine — http://clinicalresearch.med.wayne.edu/oncore.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Gardasil: Single treatment arm:
  0.5 ml single dose Gardasil vaccine given at three separate visits
  Gardasil: 0.5 ml Gardasil vaccine in single dose prefilled syringes at Visit 2, Visit 4 and Visit 6 Total of 7 study visits with vaccines given at visits 2,4 and 6
Period: Overall Study
Arm/Group | Gardasil
Started | 37
Completed | 34
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Gardasil
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 27
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Participants With Adverse Events
Description: Frequency of participants with Vaccine site reactions, Frequency of participants with Non Vaccine Adverse Events,
Time Frame: 1,61,66,181,186,211,330 days
Measure: Count of Participants; unit: Participants
Arm/Group | Gardasil
Number analyzed (Participants) | 34
Participants
  vaccine site reactions | 21
  non vaccine site reactions | 33

2. Primary Outcome: Number of Non Vaccine Adverse Events
Description: the number of non vaccine adverse events
Time Frame: 1,61,66,181,186,211,330 days
Population: Number of non vaccine adverse events
Measure: Number; unit: events
Arm/Group | Gardasil
Number analyzed (Participants) | 34
events
  non vaccine adverse events | 493
  serious adverse events | 9

3. Secondary Outcome: Seroconversion by HPV Serotypes (HPV 6, HPV 11, HPV 16, HPV 18)as Assessed by Geometric Mean Antibody Titer
Description: 1. The percentage of HPV naive women who seroconverted by HPV serotypes was measured using Geometric Mean Titers for HPV serotypes HPV 6, HPV 11, HPV 16, HPV 18
Time Frame: Baseline (prevaccine) neutralizing anti HPV antibody titers at visit 1 and anti HPV antibody titers at 1 month post 3rd vaccine shot which is at 7 months in the study.
Population: The percentage of Human Papilloma Virus (HPV) naive women for HPV serotypes 6, 11, 16 and 18 that seroconverted
Measure: Number; unit: percentage of particpants
Groups:
- HPV Serotype Naive Women: Single treatment arm:
  0.5 ml single dose Gardasil vaccine given at three separate visits
  Gardasil: 0.5 ml Gardasil vaccine in single dose prefilled syringes at Visit 2, Visit 4 and Visit 6 Total of 7 study visits with vaccines given at visits 2,4 and 6
Arm/Group | HPV Serotype Naive Women
Number analyzed (Participants) | 34
percentage of particpants
  HPV 6 Serotype: number analyzed (Participants) | 16
  HPV 6 Serotype | 100
  HPV 11 Serotype: number analyzed (Participants) | 27
  HPV 11 Serotype | 100
  HPV 16 Serotype: number analyzed (Participants) | 19
  HPV 16 Serotype | 100
  HPV 18 Serotype: number analyzed (Participants) | 27
  HPV 18 Serotype | 100

4. Secondary Outcome: SLE Disease Activity Flares
Description: SELENA-SLEDAI measurements > or = to 2 The SELENA/SLEDAI is a validated instrument which is used to score disease activity and define flares with the SELENA-SLEDAI score range being 0-105, with 0 indicating inactive disease.The SELENA/SLEDAI instrument consists of 24 items, each with a definition of activity; there are 16 clinical items and 8 laboratory items. Although there are no set standards, inactive or minimal disease is generally reflected by a SELENA/SLEDAI score of less than or equal to 2 while more than minimally active disease is reflected by a score of >2.
Time Frame: 1,61,66,181,186,211,330 days
Population: Number of patients who had a lupus flare defined by a SELENA -SLEDAI > or = to 2
Measure: Count of Participants; unit: Participants
Arm/Group | Gardasil
Number analyzed (Participants) | 34
Participants | 0

ADVERSE EVENTS:
Time Frame: Data was collected for 18 months for each patient over the trial study period
Description: Adverse events (AEs) were collected by:
  1. 30 minute post vaccine unsolicited AEs--via 30 minute post vaccine AE recording sheet
  2. 7 day post vaccine solicited AEs-- via 7 day memory aide recording sheet and reminder phone call 72 to 96 hours after each vaccination
  3. 30 day post vaccine unsolicited AEs-- via 30 day diary and weekly phone calls.
  4. weekly phone calls
  5. once per month scripted phone calls
Arm/Group | Gardasil
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 1/34
Other Adverse Events (participants affected / at risk) | 33/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gardasil (N=34)
Chest pain and arm pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Chest pain and arm pain due to atypical non cardiac chest pain and a pinched nerve affecting the arm
unplanned pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) — Unplanned pregnancy. Patient chose to terminate the pregnancy
nausea and vomiting with hypertensive crisis (Gastrointestinal disorders) | 1 (1) — Nausea and vomiting due to gastritis with dehydration Hypertensive crisis due to non compliance with hypertension medications
unplanned pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) — unplanned pregnancy. Patient chose voluntary termination of pregnancy
Chest pain and shortness of breath with left sided numbness (Musculoskeletal and connective tissue disorders) | 1 (1) — Non cardiac chest pain due to fibromyalgia. Cardiac disease ruled out.
pain, swelling and discharge of the right breast (Reproductive system and breast disorders) | 1 (1) — Pain, swelling and discharge of the right breast due to a blocked duct
shortness of breath and itching after eating peanut butter (Immune system disorders) | 1 (1) — Allergic reaction to peanut butter.Pt had known allergy to peanuts
chest pain non cardiogenic (Musculoskeletal and connective tissue disorders) | 1 (1) — Chest pain radiating down left arm due to DJD (degenerative joint disease) of the Cervical spine with radiculopathy Cardiac work up negative
swollen left leg with ulcer (Musculoskeletal and connective tissue disorders) | 1 (1) — Edema with superficial laceration which healed
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gardasil (N=34)
musculoskeletal (Musculoskeletal and connective tissue disorders) | 24 (106) — There were 106 number of musculoskeletal non vaccine related adverse events in 34 patients
nervouus system (Nervous system disorders) | 25 (106) — There were 102 Nervous system non vaccine related adverse events in 34 patients
Gastrointestinal disorders (Gastrointestinal disorders) | 18 (49) — There were 49 gastrointestinal non vaccine related adverse events in 18 patients
General disorders (General disorders) | 17 (45) — There were 45 general disorder non vaccine related adverse events in 17 patients
dermatologic (Skin and subcutaneous tissue disorders) | 17 (45) — There were 45 dermatologic non vaccine related adverse events in 17
infections (Infections and infestations) | 21 (44) — There were 44 non vaccine related infectious adverse events in 21 patients
respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 12 (29) — There were 29 respiratory non vaccine related adverse events in 12 patients
vascular disorder (Vascular disorders) | 10 (18) — There were 18 vascular disorder non vaccine related adverse events in 10 patients
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 7 (8) — There were 8 metabolism and nutrition non vaccine related adverse events in 7 patients
renal and urinary disorders (Renal and urinary disorders) | 6 (6) — There were 6 renal and urinary disorder non vaccine related adverse events in 6 people
reproductive system and breast disorders (Reproductive system and breast disorders) | 6 (7) — There were 7 reproductive and breast non vaccine related adverse events in 6 patients
psychiatric disorders (Psychiatric disorders) | 5 (12) — There were 12 psychiatric disorder non vaccine related adverse events in 5 patients
immune system disorders (Immune system disorders) | 4 (4) — There were 4 immune system disorder non vaccine related adverse events in 4 patients
Blood and Lymphatic system disorders (Blood and lymphatic system disorders) | 3 (3) — There were 3 blood and lymphatic disorder non vaccine related adverse events in 3 patients
Ear and labyrinth disorders (Ear and labyrinth disorders) | 3 (4) — There were 4 ear and labyrinth disorder non vaccine related adverse events in 3 patients
Eye disorders (Eye disorders) | 3 (3) — There were 3 eye disorder non vaccine related adverse events in 3 patients
injury poisoning and procedural complications (Injury, poisoning and procedural complications) | 3 (3) — There were 3 injury, poisoning and procedural complications in 3 patients
Surgical and medical procedures (Surgical and medical procedures) | 3 (5) — There were 5 surgical and medical procedure non vaccine related adverse events in 3 patients
Cardiac disorders (Cardiac disorders) | 2 (2) — There were 2 cardiac disorder non vaccine related adverse events in 2 patients
neoplasms benign, malignant and unspecified (incl dysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) — There were 2 neoplasms benign, malignant, and unspecified non vaccine related adverse events in 2 patients
Pregnancy , puerperium and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 2 (2) — There were 2 pregnancy, puerperium and perinatal condition non vaccine related adverse events in 2 patients
Hepatobiliary disorders-other (Hepatobiliary disorders) | 1 (1) — There was one hepatobiliary disorder non vaccine related adverse event in one patient

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No